CLINICAL TRIAL: NCT02637258
Title: Can Bedside Ultrasonographic Measurements of Optic Nerve Sheath Diameter Following the Return of Spontaneous Circulation Predict Negative Neurological Outcome in Out of Hospital Cardiac Arrest Patients?
Brief Title: Can Optic Nerve Sheath Diameter Measurement Predict Negative Neurological Outcome ?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emergency Medicine Association of Turkey (Other)
Responsible Party: Principal Investigator, Ekrem Musalar, Department of Emergency Medicine Koc University Hospital, Emergency Medicine Association of Turkey
Other Study IDs: TATDUS-0001
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Out of Hospital Cardiac Arrest; Neurologic Symptoms
Keywords: optic nerve sheath diameter; neurological outcome; OHCA
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Ultrasonographic Measurements of Optic Nerve Sheath Diameter — Bedside Ultrasonographic Measurements of Optic Nerve Sheath Diameter

SUMMARY:
This study is designed as a multicenter, prospective, cohort clinical study. The out of hospital cardiac arrest (OHCA) patients presenting to the adult emergency departments of the participating hospitals will render the study population. The non-traumatic, non-intracranial event related OHCA patients in whom the return of spontaneous circulation (ROSC) is achieved will render the sampling group.

The primary aim of this study is to evaluate the relationship of bedside ultrasound (USG) measurements of Optic Nerve Sheath Diameter (ONSD) following the ROSC after Cardiopulmonary resuscitation (CPR) for OHCA patients, with early (3rd day) neurological evaluation and 30 days survival rate, proposing that increased ONSD may be related to negative neurological outcomes. Considering a relationship is found, the secondary goals of the study are established as, identifying a cut-off value for ONSD related to negative neurological outcome and the optimal time to measure ONSD.

The sampling size with a power of 95% is calculated to be 203 patients. The patients whose available next of kin has given consent will be admitted to the study.

DETAILED DESCRIPTION:
Introduction:

Current medical literature reveals that the life expectancy after cardiopulmonary resuscitation (CPR) for out of hospital cardiac arrest (OHCA) is 6.7-9.6%.1,2 The hypoxic process, also referred to as post-resuscitation encephalopathy (PRE), is a major factor affecting the neurological outcome following return of spontaneous circulation (ROSC).3 Many studies, aiming the early prediction of the neurological outcome via vital signs, scoring systems, various biochemical markers and imaging techniques exist in literature.1-8 Optic nerve is a part of central nervous system and its posterior part is covered with dura mater. Studies have found that, elevations in intracranial pressure (ICP) resulted in elevated subarachnoid fluid pressure, leading to increased optic nerve sheath diameter (ONSD).9 Bedside USG measurements of ONSD are reported to be utilizable for evaluation of ICP.9,10

Aim of the study:

The primary aim of this study is to evaluate the relationship of bedside USG measurements of ONSD following the ROSC after CPR for OHCA patients, with early (3rd day) neurological evaluation and 30 days survival rate, proposing that increased ONSD may be related to negative neurological outcomes. Considering a relationship is found, the secondary goals of the study are established as, identifying a cut-off value for ONSD related to negative neurological outcome and the optimal time to measure ONSD.

Material and Methods:

This study is designed as a multicenter, prospective, cohort clinical study. The Utstein Templates for Resuscitation Registries are used for OHCA records.11 The associate researchers are demanded to have an experience of at least 5 years in USG use and be certified by the Emergency Medicine Association of Turkey (EMAT) for participating and/or being a faculty in the Emergency USG courses on ONSD evaluation, by the EMAT USG study group (EMATUS), which organizes planned USG courses for Emergency Physicians. A one-day education to standardize the researchers of the study, with theoretical and implementation sections are planned to be held by the authors of the study, regarding the methodology of the study and standardization of the USG techniques for ONSD measurements. In the implementation section, the researchers will perform ONSD measurements with ocular USG on healthy volunteers and the reliability among performers will be measured with Interclass Correlation test.

This study will be performed in the adult emergency departments of the participating hospitals, after the ethics committee approval. The OHCA patients presenting to the adult emergency departments of the participating hospitals will render the study population. The non-traumatic, non-intracranial event related OHCA patients in whom the ROSC is achieved will render the sampling group. The sampling size with a power of 95% is calculated to be 203 patients. The patients whose available next of kin has given consent will be admitted to the study.

All patients will receive standardized advanced cardiac life support (ACLS) measures in line with the most recent American Heart Association (AHA) guidelines by emergency department teams, uncommitted to the study. Following the ROSC, a time period of 20 minutes is determined in order to appropriate tissue perfusion to be stated, with a systolic blood pressure ≥90 mmHg or mean arterial pressure ≥65 mmHg and peripheral capillary saturation ≥94%.14 ONSD measurements will be performed in patients who had uninterrupted ROSC for 20 minutes with bedside USG and the time between the achievement of ROSC and the measurement will be recorded. The routine care plan of the patients will not be manipulated. In case the clinician decides that a cranial computed tomography (CT) is indicated according to routine practices and current guidelines, a copy of the CT images will be taken to investigate the presence of an intracranial mass leading to increased ICP.

The neurologic evaluation of the patients in the study group will be performed in three steps. Primary neurological evaluation will be performed following the achievement of appropriate tissue perfusion after ROSC, prior to any sedative or paralyzing drug application. This step is about identifying and recording the alertness, presence of activity, and the level of motor response, brain stem reflexes and myoclonic status epilepticus. The second neurological evaluation will take place after the 72nd hour following the ROSC. The alertness, presence of spontaneous motor activity, and the level of motor response, brain stem reflexes and myoclonic status epilepticus will also be identified and recorded in the second step, as well. The third evaluation will be the evaluation of neurological final outcome at 30th day or hospital discharge, utilizing the Modified Rankin Scale (MRS).

Statistical Package for the Social Sciences 22.0 for Windows will be used for statistical analysis. Descriptive statistical values will be presented as quantity and percentiles for categorical variables and as mean and standard deviation for numerical variables. Comparisons of numerical variables between two independent groups will be performed by Student-t Test if normal distribution is obtained and by Mann-Whitney U test if it is not obtained. The differences between the mean values of categorical variables of two independent groups will be tested with Chi-Square analysis. The relationships between the numerical variables will be reviewed with Pearson Correlation analysis under parametric test conditions, and Spearman Correlation Analysis under non-parametric test conditions. The appropriateness of four separately measures ONSD values will be evaluated with concordance correlation coefficient measurement. The cut-off value will be determined with Receiver Operating Characteristics Curve Analysis. The statistical alpha significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1-Out-hospital cardiac arrest

Exclusion Criteria:

1. In-hospital cardiac arrest
2. Unstable patients requiring rapid intervention (i.e. emergent surgery, percutaneous coronary intervention)
3. Age <18
4. Concomitant trauma
5. Pregnancy
6. Any event known to increase ONSD without raised ICP (optic neuritis, arachnoid cysts of optic nerve, optic nerve trauma, anterior orbital mass, cavernous sinus mass)
7. Any event known to increase ONSD with raised ICP [previously diagnosed intracranial space occupying lesion or tumor, pseudotumor cerebri, conditions causing decreased Cerebrospinal fluid (CSF) reabsorption (venous sinus thrombosis, inflammation, meningitis, subarachnoid hemorrhage)
8. Conditions causing increased production CSF (tumors), ventricular obstructions, cerebral edema, craniosynostosis
9. Anatomical eye malformations preventing the USG examination
10. Previously diagnosed malignity, glaucoma, multiple sclerosis, previously diagnosed terminal stage liver and renal disease,
11. Cardiac arrest secondary to trauma and refusing to give consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The non-traumatic, non-intracranial event related OHCA patients in whom the ROSC is achieved will render the sampling group
Sampling Method: Probability Sample
Enrollment: 203 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (MRS). | 30 day after ROSC
  0-No symptoms.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead.

SECONDARY OUTCOMES:
Neurological Examination | 72 hours after ROSC
  This step is about identifying and recording the alertness, presence of activity, and the level of motor response, brain stem reflexes and myoclonic status epilepticus.

CONTACTS AND LOCATIONS:
Overall Officials: Aslıhan Yürüktümen Ünal, Ass. Prof., Study Chair — Depertment Of Emergency Medicine, Akdeniz University, Antalya; Erkan Göksu, Ass. Prof., Study Chair — Depertment Of Emergency Medicine, Akdeniz University, Antalya; Faruk Güngör, MD, Study Chair — Depertment Of Emergency Medicine, Antalya Education and Research Hospital, Antalya; Betül Günalp, Ass. Prof, Study Chair — Depertment Of Emergency Medicine, Başkent University, Adana; Alten Oskay, MD, Study Chair — Depertment Of Emergency Medicine, Denizli State Hospital, Denizli; Mert Özen, MD, Study Chair — Depertment Of Emergency Medicine, Denizli State Hospital, Denizli; Başak Bayram, Assist. Prof, Study Chair — Depertment Of Emergency Medicine, Dokuz Eylul University, İzmir; Funda Karbek Akarca, Assist. Prof, Study Chair — Depertment Of Emergency Medicine, Ege University, İzmir; İlhan Uz, MD, Study Chair — Depertment Of Emergency Medicine, Ege University, İzmir; Nurdan Ergün Acar, Ass. Prof, Study Chair — Depertment Of Emergency Medicine, Eskisehir Osmangazi University, Eskisehir; Mustafa E. Çanakçı, Resident, Study Chair — Depertment Of Emergency Medicine, Eskisehir Osmangazi University, Eskisehir; Bülent Erbil, Ass. Prof., Study Chair — Depertment Of Emergency Medicine, Hacettepe University, Ankara; Mehmet A. Karaca, Ass. Prof., Study Chair — Depertment Of Emergency Medicine, Hacettepe University, Ankara; Özgür Dikme, MD, Study Chair — Depertment Of Emergency Medicine, Istanbul Education and Research Hospital, Istanbul; Adnan Yamanoglu, MD, Study Chair — Depertment Of Emergency Medicine, Istanbul Haseki Education and Research Hospital, Istanbul; Özgür Cevrim, MD, Study Chair — Depertment Of Emergency Medicine, Istanbul Sıslı Hamidiye Etfal Education and Research Hospital, Istanbul; Cem Ertan, Ass. Prof., Study Chair — Depertment Of Emergency Medicine, Izmır University, İzmir; Tanzer Korkmaz, Assist. Prof, Study Chair — Depertment Of Emergency Medicine, Izmır University, İzmir; Murat Yeşilaras, MD, Study Chair — Depertment Of Emergency Medicine, Izmır Tepecik Education and Research Hospital, Izmir; Turgay Y. Kılıç, MD, Study Chair — Depertment Of Emergency Medicine, Izmır Tepecik Education and Research Hospital, Izmir; Mehmet A. Aslaner, MD, Study Chair — Depertment Of Emergency Medicine, Nevşehir State Hospital, Nevşehir; Salih Ekinci, MD, Study Chair — Depertment Of Emergency Medicine, Koc University, İstanbul; Onur Karakayalı, MD, Study Chair — Depertment Of Emergency Medicine, Kocaeli Derince Education and Research Hospital, Kocaeli; Ali Batur, MD, Study Chair — Depertment Of Emergency Medicine, Erzurum Education and Research Hospital, Erzurum; Volkan Arslan, MD, Study Chair — Depertment Of Emergency Medicine, Ankara Education and Research Hospital, Ankara; Davut Kaplan, MD, Study Chair — Depertment Of Emergency Medicine, Yunus Emre State Hospital, Eskişehir
Locations (19):
- Turkey (Türkiye) (19):
  - Başkent University, Adana
  - Ankara Education and Research Hospital, Ankara
  - Hacettepe University, Ankara
  - Akdeniz University Hospital, Antalya
  - Antalya Education and Research Hospital, Antalya
  - Denizli State Hospital, Denizli
  - Erzurum Education and Research Hospital, Erzurum
  - Eskisehir Osmangazi University, Eskişehir
  - Yunus Emre State Hospital, Eskişehir
  - Istanbul Education and Research Hospital, Istanbul
  - Istanbul Haseki Education and Research Hospital, Istanbul
  - Istanbul Sıslı Hamidiye Etfal Education and Research Hospital, Istanbul
  - Koç University Hospital, Istanbul
  - Izmır University, Izmir
  - Dokuz Eylul University, Izmır
  - Ege University, Izmır
  - Izmır Tepecik Education and Research Hospital, Izmır
  - Kocaeli Derince Education and Research Hospital, Kocaeli
  - Nevşehir State Hospital, Nevşehir

REFERENCES:
- [Result] Sasson C, Rogers MA, Dahl J, Kellermann AL. Predictors of survival from out-of-hospital cardiac arrest: a systematic review and meta-analysis. Circ Cardiovasc Qual Outcomes. 2010 Jan;3(1):63-81. doi: 10.1161/CIRCOUTCOMES.109.889576. Epub 2009 Nov 10. PMID 20123673
- [Result] McNally B, Robb R, Mehta M, Vellano K, Valderrama AL, Yoon PW, Sasson C, Crouch A, Perez AB, Merritt R, Kellermann A; Centers for Disease Control and Prevention. Out-of-hospital cardiac arrest surveillance --- Cardiac Arrest Registry to Enhance Survival (CARES), United States, October 1, 2005--December 31, 2010. MMWR Surveill Summ. 2011 Jul 29;60(8):1-19. PMID 21796098
- [Result] Maramattom BV, Wijdicks EF. Postresuscitation encephalopathy. Current views, management, and prognostication. Neurologist. 2005 Jul;11(4):234-43. doi: 10.1097/01.nrl.0000159985.07242.22. PMID 15989696
- [Result] Vaahersalo J, Bendel S, Reinikainen M, Kurola J, Tiainen M, Raj R, Pettila V, Varpula T, Skrifvars MB; FINNRESUSCI Study Group. Arterial blood gas tensions after resuscitation from out-of-hospital cardiac arrest: associations with long-term neurologic outcome. Crit Care Med. 2014 Jun;42(6):1463-70. doi: 10.1097/CCM.0000000000000228. PMID 24557423
- [Result] Fugate JE, Rabinstein AA, Claassen DO, White RD, Wijdicks EF. The FOUR score predicts outcome in patients after cardiac arrest. Neurocrit Care. 2010 Oct;13(2):205-10. doi: 10.1007/s12028-010-9407-5. PMID 20645026
- [Result] Hayashida K, Nishiyama K, Suzuki M, Abe T, Orita T, Ito N, Hori S. Estimated cerebral oxyhemoglobin as a useful indicator of neuroprotection in patients with post-cardiac arrest syndrome: a prospective, multicenter observational study. Crit Care. 2014 Aug 29;18(4):500. doi: 10.1186/s13054-014-0500-6. PMID 25168063
- [Result] Daubin C, Quentin C, Allouche S, Etard O, Gaillard C, Seguin A, Valette X, Parienti JJ, Prevost F, Ramakers M, Terzi N, Charbonneau P, du Cheyron D. Serum neuron-specific enolase as predictor of outcome in comatose cardiac-arrest survivors: a prospective cohort study. BMC Cardiovasc Disord. 2011 Aug 8;11:48. doi: 10.1186/1471-2261-11-48. PMID 21824428
- [Result] Hwan Kim Y, Ho Lee J, Kun Hong C, Won Cho K, Hoon Yeo J, Ju Kang M, Weon Kim Y, Yul Lee K, Joo Kim J, Youn Hwang S. Feasibility of optic nerve sheath diameter measured on initial brain computed tomography as an early neurologic outcome predictor after cardiac arrest. Acad Emerg Med. 2014 Oct;21(10):1121-8. doi: 10.1111/acem.12477. PMID 25308135
- [Result] Hassen GW, Bruck I, Donahue J, Mason B, Sweeney B, Saab W, Weedon J, Patel N, Perry K, Matari H, Jaiswal R, Kalantari H. Accuracy of optic nerve sheath diameter measurement by emergency physicians using bedside ultrasound. J Emerg Med. 2015 Apr;48(4):450-7. doi: 10.1016/j.jemermed.2014.09.060. Epub 2014 Dec 9. PMID 25497897
- [Result] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900
- See also: Standardized echography of the optic nerve — http://link.springer.com/chapter/10.1007%2F978-94-011-1846-0_1#page-1
- See also: Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A consensus statement from the International Liaison Committee on Resuscitation — http://www.ncbi.nlm.nih.gov/pubmed/?term=18948368
- See also: Utstein Collaborators — http://www.ncbi.nlm.nih.gov/pubmed/?term=25438254